CLINICAL TRIAL: NCT06229691
Title: Muscle Fatigability and Trip-specific Fall Risk in Adults With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1924071; U54GM104941 (NIH)
Record Dates: First submitted 2024-01-05; First posted 2024-01-29 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Osteoarthritis, Knee
Keywords: balance; fatigue; falls
MeSH Terms: conditions — Osteoarthritis, Knee; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy (Experimental)
  Interventions: Behavioral: 30 minute treadmill walk
- Knee osteoarthritis (Experimental)
  Interventions: Behavioral: 30 minute treadmill walk

INTERVENTIONS:
Behavioral: 30 minute treadmill walk — Participants will walk on a treadmill at their preferred speed for 30 minutes. One minute "challenge" periods will occur at minutes 7, 17, and 27, when the treadmill speed will increase by 50%. This walk will induce a magnitude of muscle fatigue corresponding to an individual participant's fatigability.

SUMMARY:
The goal of this clinical trial is to learn about how fatigue affects the risk of falling in adults aged 55-70 years with and without knee osteoarthritis. The main questions this trial aims to answer are:

* Does fatigue increase the risk of tripping while walking? and
* Does fatigue increase the risk of falling in response to a trip while walking? Participants will
* Complete questionnaires
* Wear a device that measures physical activity for 5-7 days
* Complete a 30 minute walk on a treadmill
* Complete the following before and after the treadmill walk:

  * Computer test to measure mental fatigue
  * Maximal strength testing
  * Balance test

Researchers will compare adults with and without knee osteoarthritis to see if fall risk in adults with knee osteoarthritis is affected more by walking activity compared to adults without knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

For adults with knee osteoarthritis:

* presence of occasional to frequent knee pain
* knee pain that is primarily in the medial knee joint compartment
* minimal morning joint stiffness

For all participants:

* able to walk continuously for 30 minutes without an assistive device

Exclusion Criteria:

* fracture or surgery within 1 year
* history of joint replacement
* lower-extremity joint injections within 3 months
* history of stroke or other neurological condition
* cardiovascular or pulmonary conditions that limit daily activity or that preclude participation in exercise
* history of major lower extremity or back injury or pain (except for knee osteoarthritis)
* history of lower extremity amputation
* use an orthotic or prosthetic to walk
* use of beta blockers or other medications that affect fatigue
* use of medications that affect balance
* diabetic neuropathy
* acute illness or the presence of lesions on the torso or lower extremities
* BMI greater than 35
* body weight over 265 lbs

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-05-14 (Actual); Primary Completion 2025-08-27 (Actual); Study Completion 2025-08-27 (Actual)

PRIMARY OUTCOMES:
Minimum toe clearance during walking | Beginning and end of 30 minute treadmill walk
  Minimum toe clearance will be calculated from the first and last minutes of the treadmill walk using optical motion capture.
Anterior stability margins during walking | Beginning and end of 30 minute treadmill walk
  Anterior stability margins will be calculated from the first and last minutes of the treadmill walk using optical motion capture.
Anterior reactive stepping | Beginning and end of 30 minute treadmill walk
  Stability margins will be calculated from a lean-release test conducted before and after the 30 minute treadmill walk
Knee extensor fatigability | Before and after the 30 minute treadmill walk
  Knee extensor fatigability will be calculated as the change in maximum knee extensor power (measured via dynamometry) pre- to post-30 minute treadmill walk

CONTACTS AND LOCATIONS:
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No